CLINICAL TRIAL: NCT03786510
Title: A Pilot Study on the Effectiveness of Multidomain Intervention Program for Reducing Risks of Dementia
Brief Title: A Study on the Effectiveness of Multidomain Intervention Program for Reducing Risks of Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul Metropolitan Government (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MDP_AD
Record Dates: First submitted 2018-12-17; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Alzheimer Disease
Keywords: Risk reduction; Community; Older adults; Lifestyle modification
MeSH Terms: conditions — Alzheimer Disease; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: A single-blinded randomized controlled pilot study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active control (Active Comparator): The control group received Community Center for Dementia's usual care of regular health check-up.
  Interventions: Behavioral: Active control
- Intensive + Maintenance program (Experimental): The INT+MNT group participated in a 4-week intensive program followed by a 20-week maintenance program
  Interventions: Behavioral: Intensive + Maintenance program
- Intensive program only (Experimental): The INT only group participated in a 4-week intensive program
  Interventions: Behavioral: Intensive program only

INTERVENTIONS:
Behavioral: Active control — Control group received a personalized advice on lifestyle modification to prevent dementia and usual care of Community Center for Dementia.
  Arms: Active control
Behavioral: Intensive + Maintenance program — Both intensive and maintenance program
  1. Intensive program The 4-week group-based intensive program was comprised of eight sessions; each session consisted of (1) a 30-min review of the tasks, (2) a 50-min training period, and (3) a 10-min meeting to assign tasks on an individual basis. A study nurse-guided training for modification of vascular risk factors, diet, cognitive and social activity were conducted, And, a physiotherapist conducted an exercise training mainly composed of muscle strengthening and stretching.
  2. Maintenance program The allocated study assistants monthly check-up whether participants adhere to the altered habits or not, based on the workbook
  Arms: Intensive + Maintenance program
Behavioral: Intensive program only — Only the intensive program was conducted.
  The 4-week group-based intensive program was comprised of eight sessions; each session consisted of (1) a 30-min review of the tasks, (2) a 50-min training period, and (3) a 10-min meeting to assign tasks on an individual basis. A study nurse-guided training for modification of vascular risk factors, diet, cognitive and social activity were conducted, And, a physiotherapist conducted an exercise training mainly composed of muscle strengthening and stretching.
  Arms: Intensive program only

SUMMARY:
Investigators aimed to examine the feasibility and effectiveness of a multidomain intervention strategy involving intensive and maintenance programs aimed at reducing the risk of Alzheimer's disease (AD) in at-risk older adults. Participants were randomly allocated into three groups: (1) intensive plus maintenance program (INT+MNT group), (2) intensive program only (INT-only group), and (3) active control (control group). There were two study hypotheses: 1) the participants in the 4-week intensive program (INT+MNT and INT-only group) would show reduced dementia risk scores compared to control; and 2) that the participants in the added 20-week maintenance program (INT+MNT group) would show greater improvement in dementia risk scores compared to the INT-only and control groups.

DETAILED DESCRIPTION:
OBJECTIVES: To examine the feasibility and effectiveness of a multidomain intervention strategy involving intensive and maintenance programs aimed at reducing the risk of Alzheimer's disease (AD) in at-risk older adults.

DESIGN: A prospective randomized controlled trial with participants assigned to three parallel programs: intensive plus maintenance (INT+MNT), intensive only (INT-only), and active control.

SETTING: A community center for dementia in South Korea.

PARTICIPANTS: Community-dwelling older adults (aged ≥ 60 years) without dementia, but having several risk factors for AD.

MEASUREMENTS: The study subjects participated in a 4-week intensive group-based lifestyle modification program that focused on physical activity, vascular risk factors, dietary habits, cognitive activities, and social engagement. Then, the participants underwent a 20-week maintenance program to consolidate modified habits. Linear mixed models were used to examine the changes in modified Australian National University-Alzheimer's Disease Risk Index (ANU-ADRI) scores in each group. Additional analyses of secondary outcomes, including cognitive function, were also performed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 60 years and over with age-, sex-, education-adjusted z-score of the Korean version of mini-mental state examination for dementia screening (MMSE-DS) -1.5 standard deviation and above, but having some risk factors for dementia were included: at least two of following risk factors in a recent year (1) do not exercise with moderate degree more than 3 times a week, (2) do not read books, newspapers or magazine more than once a week; (3) do not meet friends, relatives, or close person more than once a week, (4) have depressed mood or low volition.

Exclusion Criteria:

* Exclusion criteria were previously diagnosed with dementia or other neurologic disorders (e.g., Parkinson's disease); stroke in a recent year or having significant sequelae of past stroke; major psychiatric disorders (e.g., major depressive disorder) in a recent year; having absolute contraindication to participate in exercise program (e.g., need a wheelchair for mobility). Also, subjects who were already participated in other exercise or cognitive stimulating program in the Community Center for Dementia were excluded in the present study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline Australian National University Alzheimer's Disease Index (ANU-ADRI) at 4 weeks and 24 week | baseline (0 week), 4-week, 24-week
  The ANU-ADRI was developed based on review and meta-analysis of the literature regarding modifiable risk and protective factors for AD; it is a validated instrument assessing individual risk profiles for AD that combines the odds ratios of risk factors to derive a risk score. The total scores ranged from -18 to 63 for males, and from -18 to 66 for females; higher scores indicated greater risk for AD.

SECONDARY OUTCOMES:
Changes from baseline Short Physical Performance Battery (SPPB) at 4 weeks and 24 week | baseline (0 week), 4-week, 24-week
  The SPPB was developed for evaluating lower extremity functioning in older persons. The scores range from 0 to 12; higher scores indicated better performance.
Changes from baseline total score in the CERAD neuropsychological battery at 4 weeks and 24 week | baseline (0 week), 4-week, 24-week
  The CERAD neuropsychological battery includes various cognitive domains: memory, language, visuospatial, executive, etc. There are age-, sex-, and educational year-stratified norms; individuals' z-score can be calculated.
Changes from baseline Color Word Stroop Test (CWST) at 4 weeks and 24 week | baseline (0 week), 4-week, 24-week
  CWST mainly can examine the executive function. There are age-, sex-, and educational year-stratified norms; individuals' z-score can be calculated.
Changes from baseline Seoul-Instrumental Activities of Daily Living (S-IADL) at 4 weeks and 24 week | baseline (0 week), 4-week, 24-week
  The S-IADL includes 15 items in regard with various instrumental activities of daily living. The total scores ranged from 0 to 15; higher scores indicated lower level of daily function.
Changes from baseline EuroQol Five-Dimensional Questionnaire (EQ-5D) at 4 weeks and 24 week | baseline (0 week), 4-week, 24-week
  The EQ-5D is consisted of five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The total scores ranged from 5 to 15; higher scores indicated lower quality of life.
Changes from baseline Motivation to Change Lifestyle and Health Behaviors for Dementia Risk Reduction Scale (MCLHB-DRR) scale at 4 weeks and 24 week | baseline (0 week), 4-week, 24-week
  The MCLHB-DRR was developed to understand beliefs underpinning the lifestyle and health behavioural changes needed for dementia risk reduction. Seven-factor solution (perceived susceptibility, perceived severity, perceived benefits, perceived barriers, cues to action, general health motivation, self-efficiency) with 27 items were included. The total scores ranged from 0 to 27; higher scores indicate higher motivation for reducing risk of dementia

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided